CLINICAL TRIAL: NCT03871907
Title: Effect of Digital Technologies on Risk Factor Modification in Patients After Percutaneous
Brief Title: Effect of Digital Technologies on Risk Factor Modification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DigTech
Record Dates: First submitted 2019-03-06; First posted 2019-03-12 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Digital Technology

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigators who will perform follow-up will be masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital technology (Active Comparator): standard cardiac rehabilitation program + 4 personalized short messages about risk factors modification 4 times per week
  Interventions: Behavioral: Digital technology
- Control (No Intervention): standard cardiac rehabilitation program

INTERVENTIONS:
Behavioral: Digital technology — Lifestyle-Focused Text Messaging
  Arms: Digital technology

SUMMARY:
DigTech investigates the effect of a text message-based intervention to encourage lifestyle change on objective measures of cardiovascular risk in individuals with coronary heart disease (CHD) after percutaneous coronary intervention (PCI).

DigTech will recruit 700 participants from 18-75 years old with CHD after PCI. Half of the participants will be randomised into a 24 week intervention trial, which includes sending 4 personalized short messages about risk factors modification 4 times per week and the other half will be controls.

Participants will complete 3 main study visits:

* Visit 1: Baseline visit conducted at the beginning of the study
* Visit 2: Randomization
* Visit 3: End of study (24 weeks). Each visit will repeat the same set of cardiovascular measures including information about previous treatment, blood pressure, ECG, echocardiography, stress tests, blood sampling, International Physical Activity Questionnaires (IPAQ) and other measures.

DETAILED DESCRIPTION:
DESIGN: DigTech is a parallel-group, single-blind, randomized clinical trial investigating the changes in cardiovascular risk factors (low-density lipoprotein cholesterol [LDL-C] level, blood pressure, body mass index [BMI]) according to personalized intervention, based on individual short messages in CHD patients after PCI.

BACKGROUND AND AIMS:

Cardiovascular disease prevention, including lifestyle modification, is important but underutilized. Mobile health strategies could address this gap but lack evidence of therapeutic benefit.

This trial aims at the examination of the effect of a lifestyle-focused personalized support program delivered by mobile phone text message on cardiovascular risk factors.

PARTICIPANTS: 700 participants aged 18-75 with CHD after PCI.

RECRUITMENT: Tyumen Cardiology Research Center, branch of the Tomsk NRMC

CONFIDENTIALITY: All information and documents collected will be stored securely and kept in strict confidence in compliance with regulatory acts.

Study samples, investigation results and incidental findings. The use of the participants' study samples and investigations are clearly defined in the participant information leaflet and will be explained during the informed consent process.

CONSIDERATION OF NULL HYPOTHESES: A null hypotheses that personalized lifestyle intervention based on received 4 text messages per week for 6 months in addition to usual care in CHD patients after PCI does not reduce LDL-C levels, blood pressure and BMI" was not selected.

SAMPLE SIZE SELECTION: Prior study shows that a sample size of 634, increasing to 704 to allow for a10% loss to follow-up, would have 90% power (2-tailed and at a 5% significance level) to detect a difference of 10 mg/dL in LDL-C level.

INTERVENTION: The text message will be based on the prevention program involved delivery of regular personalized text messages (some messages personally addressed through a "mail-merge"-type function with the participant's preferred name) providing advice, motivation, and information that is aimed to improve diet, increase physical activity, and encourage smoking cessation (if relevant). Content for each participant will be selected using a re-specified algorithm dependent on key baseline characteristics. Participants will receive 4 messages per week for 24 weeks. Each message will be sent on 4 of 5 randomly selected days and arrived at random times of the day during working hours. The content of messages will be based on national guidelines on cardiovascular disease prevention.

STUDY PROCEDURES AND DATA COLLECTION

SCREENING VISITS: Screening Visit Procedures (Visit 0). Evaluation of inclusion and exclusion criteria. Patients will provide written informed consent on this visit.

MAIN STUDY VISITS COMPLETION OF STUDY VISITS 1-3

There are three main visits planned for each participant:

Visit 1: conducted at the beginning of trial (baseline).

* Questionnaire. It will collect detailed information about physical activities (International Physical Activity Questionnaires short form) and also lifestyle information such as daily routines and use of alcohol and tobacco, information about previous treatment.
* Physical Measures. Investigators will measure blood pressure, height, weight, BMI, heart rate.
* Cardiovascular Measures:

  1. Electrocardiogram (ECG).
  2. Echocardiogram
  3. Six Minute Walk Test.
  4. Coronary angiography
* Blood Sampling including blood lipid spectrum (total cholesterol, triglycerides, cholesterol high-density lipoproteins and cholesterol low-density lipoproteins). Fasting blood samples will be analyzed by local laboratories.

Visit 2: Randomization. Randomization will be performed after PCI, prior to discharge from the hospital.

Randomization will occur via a computerized randomization program that will access through a secure web interface. The random allocation sequence will be in a uniform 1:1 and will be concealed from study personnel. Study staff will enroll patients by entering data into the secure web interface. The computerized randomization program interfaced with the message-sending program to trigger the sending of messages to patients randomized to the intervention. To maintain blinding of personnel study, patients will be informed of their allocation in a text message sent after hospital discharge. Prior to their follow-up appointment patients also will receive a text message to ask them not to reveal their allocation status to study personnel or clinicians in follow-up visits. Intervention participants will receive, in addition to usual care, the 6-months prevention program of approximately 96 messages. Control participants will receive usual care, which generally included community follow-up with the majority referred to inpatient cardiac rehabilitation, as determined by their usual physicians.

Visit 3: conducted after 24 weeks (at the end of the trial, Follow-up visit).

ANALYSIS: Patient demographic characteristics and other baseline information will be summarised by treatment group. Numbers (with percentages) for binary and categorical variables and mean (standard deviation), or median (interquartile or full range) for continuous variables will be presented. Normality of variables will be assessed by visual assessment of the normality curves and the Kolmogorov-Smirnov test. The analysis of the primary outcome will be assessed using analysis of covariance (ANCOVA) adjusting for baseline values and minimisation factors used in the randomisation process. Results will be presented as adjusted mean difference in change in ambulatory blood pressure between randomised groups at 4 months with 95% confidence intervals (CI) and associated two-sided p value. The above method was also used for continuous secondary outcomes. With respect to management of combined risk factors, the proportion of patients achieving control of risk factors was analyzed in terms of relative risk at month 6 and compared between groups using a log-binomial regression. If the model assumptions are not met and evidence of departure from Normality is observed, transformations of the data will be employed or non-parametric tests will be carried out. Statistical analysis will be carried out using SPSS statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease at the age of 18 to 75 years who are planning PCI for hemodynamically significant coronary artery stenosis.

Exclusion Criteria:

* Severe comorbidities (malignant tumors, severe lung diseases, marked cognitive impairment).
* Severe CHF (EF LV <35% or functional class of heart failure III-IV NYHA).
* Severe valvular heart disease or Prosthetic heart valves.
* Severe diseases of the musculoskeletal system.
* The patient's reluctance to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Low-density lipoprotein cholesterol level at 6 months | 6 months
  The primary end point was low-density lipoprotein cholesterol level at 6 months

SECONDARY OUTCOMES:
Systolic blood pressure | 6 months
  Systolic blood pressure will be lower in the intervention group compared with the control group
Body mass index (BMI) | 6 months
  Body mass index (weight and height will be combined to report BMI in kg/m^2) will be lower in the intervention group compared with the control group

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V Popov, Principal Investigator — Tomsk National Research Medical Center of the Russian Academy of Sciences
Locations (1):
- Tyumen Cardiology Research Center, Tomsk National Research Medical Center, Russian Academy of Science, Tyumen, Russia

IPD SHARING:
Plan to Share IPD: No